CLINICAL TRIAL: NCT06414057
Title: HPV Equity Study: Exploring Cervical Cancer Control in Scotland for Women With Experience of Priority Risks
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC23210
Record Dates: First submitted 2024-05-10; First posted 2024-05-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Human Papilloma Virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal swab for HPV genotyping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Investigators will offer Gardasil-9 and HPV self-swab screening to up to 500 individuals across the three study sites, aiming to recruit 120-180 individuals within each of the three participating health boards over a 6-9 month timeframe. Participants will be asked to provide a vaginal swab sample for baseline HPV testing.
  Interventions: Other: Offering opportunistic HPV vaccine during routine sexual health clinic visits

INTERVENTIONS:
Other: Offering opportunistic HPV vaccine during routine sexual health clinic visits — Investigators will offer Gardasil-9 and HPV self-swab screening to up to 500 individuals across the three study sites, aiming to recruit 120-180 individuals within each of the three participating health boards over a 6-9 month timeframe. Participants will be asked to provide a vaginal swab sample for baseline HPV testing.

SUMMARY:
Individuals with experience of homelessness, substance use/addiction, transactional sex, and incarceration experience significant health inequities across a wide range of health conditions. This inequity includes cervical cancer with individuals in these populations less engaged with both routine human papillomavirus (HPV) vaccination and cervical cancer screening programmes, yet also at higher risk of developing cervical cancer.

Opportunistic vaccination is recommended by the Joint Committee on Vaccination and Immunisation for 'other at risk/vulnerable groups' who may benefit (such as people with experience of transactional sex or incarceration) at clinical discretion. However, there is limited evidence on the feasibility, uptake, attitudes and impact of vaccination in these at-risk groups and no nationally funded programme.

This mixed methods exploratory study seeks to generate evidence to inform the optimal service design. Core objectives are to: 1) assess the feasibility and acceptability of offering opportunistic HPV vaccination during standard sexual health care to women at high risk of HPV and cervical cancer; 2) identify the type-specific prevalence of HPV among recruited participants; and 3) describe participants' perceptions and experiences of accessing routine HPV vaccination and cervical screening services, and/or this opportunistic (research) service.

The investigators will seek to recruit women with experience of homelessness, substance use/addiction, transactional sex, and incarceration. The study will include trans-men and non-binary people at risk of cervical cancer with the same risk experiences. Potential participants will be identified prospectively via attendance at specialist sexual health services in Scotland.

Participants will be offered HPV vaccination and testing, and/or an in-depth research interview. Participation can be completed within one clinic visit. The full vaccination course is available via participation (min/max does spacing 6/12 months) and participants testing positive for high-risk type HPV can/will be followed up in full and supported in accessing treatment.

DETAILED DESCRIPTION:
Component 1: Focusses on assessment of the prevalence of HPV in our study population, and on the provision, and assessment of the uptake, of HPV vaccination (gardesil-9).

Intervention - HPV vaccination and self-swab screening will be offered to up to 500 individuals across the three study sites, aiming to recruit 120-180 individuals within each of the three participating health boards over a 6-9 month timeframe.

Vaccine provision - All aspects of the vaccine provision in this study will be conducted in line with current clinical practice and follow the site's local GPD for HPV vaccine provision. The cost of vaccine provision in this study is being met by charitable donation of the standard vaccine by the pharmaceutical company (MSD).

Vaccine - This study will use Gardasil-9, produced and provided by MSD. It is a nine valent vaccine offering protection against HPV types 6, 11, 16, 18, 31, 33, 45, 52 & 58, and is the only vaccine available to use in the UK.

Number of doses - The risk profile of the participant population is considered to be similar to that of GBMSM. Accordingly, participants will be offered 2/3 doses of the vaccine according to their immunocompetency.

HPV testing - Participants will be asked to provide a baseline self-taken vaginal swab for HPV testing. Self-swab sampling is being offered as this is standard practice for Chlamydia and Gonorrhoea testing, increasing uptake for individuals who would decline an examination, such as those with experience of sexual trauma. If participants would rather not take a self-taken swab, then clinician taken sampling will be offered.

Swab tests - This study will use the COPAN FloqSwabs™; pictorial instructions for sampling will be provided. Swabs will be dispatched to the Scottish HPV Reference Laboratory (SHPVRL) for HPV genotyping.

Laboratory analysis - HPV genotyping will be performed using the AllplexT HPV 28 assay.

Follow-up of HPV+ participants - All participants with a positive high-risk type HPV test on their swab will be contacted and advised that a liquid-based cytology (LBC) smear test is recommended.

Travel expenses - Participants will be offered travel expenses (up to £25 in total) for attendance at the clinic for repeat vaccine doses or follow-up smear test.

-----------------------------------

Component 2: consists of a qualitative exploration of the perspectives of women from our target population on HPV vaccination and screening.

In-depth interview study - Investigators will conduct individual interviews with people invited to take part in the vaccine intervention study. This will include individuals who accepted the vaccine and screening and those who declined.

Recruitment - Participants will be invited to consider taking part in a research interview at the same time as recruitment to component 1. This will include individuals who choose to undertake the vaginal sampling and HPV vaccination, or after refusing to do so. It will be made clear that this is an additional, optional, component and that the interview would be carried out by a University of Edinburgh researcher, and will be held a safe environment.

Up to 30 interviews will be conducted across the three health boards, seeking to include a balance of participants from each of the eligible groups. Participants will be offered a £10 voucher in recognition of their time. The voucher will only be given following the completion of the interview. For participants currently living in custody, £10 will be added to their commissary account.

Interview conduct - Interviews will be carried out by an experienced researcher and will explore topics related to cervical cancer/HPV risks, vaccination, and access to current vaccine and cervical screening services. Interviews will take a semi-structured format and the interviewer will be free to pursue any relevant line of conversation appearing to be of importance to that participant.

Interviews will be carried out in a private space in person (in either the clinic facility/outreach facility) or via phone, or via the approved NHS digital remote consultation platform if the participant is currently in prison. Interviews will be recorded on an encrypted device and transcribed verbatim. Investigators will use a university approved company (First Class Secretarial Services) with a confidentiality and data-processing agreement in place, and transcripts will be checked for accuracy and fully anonymised by the Lead Research Fellow.

Analysis - analysis will be undertaken using an abductive thematic approach (i.e. we will look for patterns, themes, and connections in participants' accounts. Investigators will commence coding and analysis with an outline codebook based on relevant established literature and theories, and will use new insights and perspectives gained directly from the data to add new codes and adapt the coding structure during the analytical process).

The NVivo software (QSR NVivo version 10) will be used to store and organise the transcripts, and all coding and analysis undertaken.

Interpretation - Individual member checking may be challenging for some participants however, PPI input to the interpretation and reporting of interview findings will be obtained from the study advisory panel which will include representatives from advocacy groups such as Jo's Cervical Cancer Trust, and the Waverly Centre. Where appropriate, the Research Fellow will attend advocacy groups to ensure participant group views are suitably represented in the interpretation of the results.

ELIGIBILITY:
Inclusion Criteria:

Individuals will be eligible for participation in components 1 and/or 2 if they:

* have a cervix
* are aged 25-45 years (inclusive)
* are able to provide informed consent for themself

And have experience of either:

* substance use/addiction
* living in custodial settings
* homelessness
* involvement in transactional sex

Exclusion Criteria:

Individuals will be excluded from participation if they:

* Do not have a cervix due to surgery or other reasons
* Are known to have completed the full vaccination schedule (as per JCVI criteria for their age and immunocompetency) (Excluded from component 1 (vaccination and HPV screening) only - still able to participate in component 2 (individual interview))
* Meet any of the vaccine exclusion criteria as set out in the local HPV PGD
* Have had a confirmed anaphylactic reaction to a previous dose of HPV vaccine.
* Have had a confirmed anaphylactic reaction to any component of the vaccine. Practitioners must check the marketing authorisation holder's SmPC for details of vaccine components.
* Have a history of severe (i.e. anaphylactic reaction) to latex where the vaccine is not latex free.
* Are known to be pregnant.
* Are suffering from an acute severe febrile illness (the presence of a minor infection is not a contraindication for immunisation).

Additionally, PGDs advise caution where a neurological condition is believed to be progressing or there is neurological deterioration and therefore, individuals meeting this criteria will be excluded (from component 1 only).

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult women, trans men, or non-binery individuals with a cervix attending routine sexual health services who aslo have experience of substance use/addiction, living in custodial settings, homelessness, or involvement in transactional sex.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Uptake | Baseline
  Number of participants taking up HPV screening and initial HPV vaccine dose during the clinic visit

SECONDARY OUTCOMES:
Clinician/self sampling | Baseline
  Proportion of participants who provide a self-taken vaginal swap/opt for a clinician-taken swab
Vaccine completion | 12 months
  Number of participants completing vaccine schedule, assessed in line with JCVI guidance
HPV prevalence | 4 weeks
  Number of participants testing HPV + for each sub-type
Follow-up tests | 6 months
  Number of participants undertaking clinical follow-up after testing HPV + for high risk variant

CONTACTS AND LOCATIONS:
Overall Officials: Christine Campbell, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be made available as we will be undertaking a follow-up study in 5-10 years